CLINICAL TRIAL: NCT00040131
Title: Safety and Efficacy Study of IL-10 (Tenovil TM) in the Prevention of Post-ERCP Acute Pancreatitis (Study P02580)(TERMINATED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: P02580
Record Dates: First submitted 2002-06-20; First posted 2002-06-21 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Bile Duct Diseases; Biliary Tract Diseases; Gallbladder Diseases; Pancreatitis; Pancreatic Diseases
MeSH Terms: conditions — Bile Duct Diseases; Biliary Tract Diseases; Gallbladder Diseases; Pancreatitis; Pancreatic Diseases | interventions — Interleukin-10

INTERVENTIONS:
Drug: IL-10

SUMMARY:
The purpose of this study is to determine if a single dose of IL-10 compared to placebo is safe and effective in reducing the incidence of post-ERCP acute pancreatitis for subjects with increased risk.

ELIGIBILITY:
Inclusion criteria:

Adults weighing up to 125 kg who are undergoing ERCP for any of the following:

* Evaluate recurrent abdominal pain;
* Evaluate unexplained recurrent pancreatitis;
* Evaluate prior post-ERCP pancreatitis;
* Treatment of pancreatic disorders;
* Treatment of Common Bile Duct Stones (without jaundice)

Exclusion criteria:

* Active (acute) pancreatitis;
* Chronic pancreatitis (moderate and severe cases);
* ERCP to perform a second procedure on biliary tract;
* Patients who previously had pancreatic sphincterotomy;
* Known or suspected pancreatic cancer or cancer of Papilla of Vater;
* Known or suspected other malignancy;
* History of, or current clotting or bleeding problems;
* Moderate and severe Anemia;
* Low platelet counts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2002-01; Primary Completion 2002-12 (Actual); Study Completion 2003-01 (Actual)